CLINICAL TRIAL: NCT02893943
Title: Impact of Probiotics on Weight Control and Body Composition in Overweight and Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2016:033
Record Dates: First submitted 2016-08-29; First posted 2016-09-09 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Probiotics (Active Comparator): 1 capsule per day containing probiotics
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): 1 capsule per day without probiotics
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the potential of probiotics on weight management. It is hypothesized that the consumption of 1 capsule of probiotics daily will modulate the intestinal gut microbiota thereby reducing body weight and fat compared to those who do not consume probiotics. In addition, a diet supplemented with probiotics can be expected to be more beneficial than a diet without probiotic supplementation in impacting biomarkers of obesity-associated disorders including diabetes, hypertension and cardiovascular disease (CVD).

DETAILED DESCRIPTION:
Overweight, obese men and women volunteers aged between 18-65 yrs with BMI greater than or equal to 25 will be recruited from the Winnipeg (Manitoba, Canada) area to participate in a two arm crossover, randomized, double-blind, placebo-controlled, free-living intervention study for 60 days per study period following obtainment of informed consent. Participants will be informed to maintain their usual diets as well as their physical activity level.

After obtaining consent, participants will be randomized to receive either 1 capsule containing probiotics, or 1 capsule of placebo daily for 60 days. Compared with the probiotic capsules, the placebo contains the same carrier material and is similar in size, shape and taste.

ELIGIBILITY:
Inclusion Criteria:

* Overweight, obese men and women volunteers aged between 18-65 yrs
* BMI equal to or greater than 25
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits.
* Willingness to discontinue consumption of fermented foods or probiotics (e.g. yoghourts, with live, active cultures or supplements), laxatives, prebiotics and any substances for control body weight.
* Able to provide informed consent.
* Women of childbearing potential with a negative pregnancy test at screening.

Exclusion Criteria

* BMI greater than 35
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorptive syndrome, pancreatitis, gallbladder or biliary disease.
* Those currently taking (or have taken within the last 3 months) cholesterol-lowering, triglyceride-lowering or hypertension medications.
* Those currently taking (or have taken within the last 3 months) lipid-lowering supplements, (e.g., omega-3 supplements, plant sterols/stanols foods and/or supplements, fibre, etc).
* Smokers.
* Allergic to milk, soy, or yeast (some of our probiotics strains may contains these items).
* Use of another investigational product within 3 months of the screening visit.
* Positive pregnancy test in women of child-bearing potential.
* Known to be pregnant or breast-feeding or planning on becoming pregnant in the next 18 months.
* Women of child-bearing potential not using effective contraception.
* Use of any other treatments (medication or nutritional program) affecting body weight, food intake and/or energy expenditure.
* Menopausal women.
* Weight gain or loss of at least 10lbs in previous three months.
* Uncontrolled angina within the past six months.
* Cancer treatment (radiation, chemotherapy, surgery) within past six months or any other treatment or condition known to weaken the immune system (such as systemic corticosteroids or HIV/AIDS).
* Any physical condition deemed likely to significantly interfere with individuals' ability to participate in a nutritional intervention.
* Currently or at any point during the study participating in Weight Watcher's or another weight loss program or taking a medication for weight loss.
* History of drug or alcohol (> 2 drinks daily) abuse.
* Abnormal thyroid hormone levels.
* Immune-compromised conditions.
* Participant experiencing nausea, fever, vomiting, bloody diarrhoea or severe abdominal pain (past week and chronic).
* Participants exercising > 15 miles/wk or 4,000 kcal/wk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Body weight | 60 days

SECONDARY OUTCOMES:
Body mass index | 60 days
Body fat percentage | 60 days
Waist circumference | 60 days
Hip circumference | 60 days
Total fat mass | 60 days
Total lean mass | 60 days
Gut microbiome | 60 days
  Stool samples will be collected from participants to analyze intestinal microbiota community composition
Blood pressure | 60 days
Blood total cholesterol | 60 days
Blood low-density lipoprotein cholesterol | 60 days
Blood high-density lipoprotein cholesterol | 60 days
Blood triglycerides | 60 days
Blood glucose | 60 days
Blood insulin | 60 days
Aspartate aminotransferase | 60 days
Alanine transaminase | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Rotimi Aluko, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada